CLINICAL TRIAL: NCT03259139
Title: Effect of Exposure to Gun Violence in Video Games on Children's Interest in Real Guns: A Randomized Clinical Trial
Brief Title: Exposure to Gun Violence in Video Games Increases Interest in Real Guns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Brad Bushman, Professor of Communication & Psychology, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 2013B0542
Record Dates: First submitted 2017-07-22; First posted 2017-08-23 (Actual); Results first posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: Psychology, Social; Adolescent Behavior
Keywords: adolescent; gun; violence; media
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to play a non-violent video game, a violent video game containing swords, or a violent video game containing guns.
Who Masked: Participant
Masking Description: Participants did not know which condition they were in. Participants' parents were aware of the deception (hidden guns) and what condition their children were in. Research personnel knew conditions as well. Research assistants who transcribed recorded laboratory sessions did not know what condition they were coding (eg. what type of game they played)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Violence with guns (Experimental): Participants in this condition will play a video game with violent content which includes guns.
  Interventions: Behavioral: Video games and violence
- Experimental: Violence without guns (Experimental): Participants in this condition will play a video game with violent content which does not include guns. Instead, the violence will include weapons such as swords.
  Interventions: Behavioral: Video games and violence
- Control: No violence (Other): Participants in this condition will play a video game which contains no violent content or weapons.
  Interventions: Behavioral: Video games and violence

INTERVENTIONS:
Behavioral: Video games and violence — Participants will be randomly assigned to play a video game which contains either (1) no violent content, (2) violent content with swords, or (3) violent content with guns. The game, rated E, is age appropriate and modded to include guns in the appropriate condition.

SUMMARY:
More American children die by accidental gun use than children in other developed countries. One factor that can influence children's interest in guns is exposure to media containing guns. The objective of this study is to test whether children who play a video game containing guns will handle a real gun longer, will pull the trigger more times, and pull the trigger while pointing the gun at themselves or another than children who see the same movie without guns.

DETAILED DESCRIPTION:
The design will be a 2 (player vs. observer) x 3 (nonviolent, violent with sword, violent with gun) between-subjects study. Participants will randomly be assigned to conditions. Participants will be tested in pairs. The participant in the player condition will play a video game while the participant in the watcher condition will watch. The participants will be in the same room, seated next to each other.

Video games will be chosen for the three conditions which have no violent content (nonviolent condition), violent content with a sword as a weapon for the player (violent with sword condition), and violent content with a gun as a weapon (violent with gun condition). All games chosen will be age appropriate (rated E) and have a consistent perspective (i.e., 1st person or 3rd person) between conditions. Participants will be asked how familiar they are with the video game used to control for experience with the stimulus. Gameplay will last for 20 minutes.

The measures for experiment 3 will include the media habits, aggressive behavior, attitude toward guns, and guns in the home measures listed for experiment 1. In addition, parents will be asked if their children have taken a gun safety course and a behavioral measure will be whether or not children handle a real (but non-firing) gun and whether they pull the trigger.

Participants will be tested in pairs, with a sibling or friend. Participants will be placed in a room containing toys, with a camera on the wall. Participants will be told that they can play with any of the toys in the room for the next 20 minutes. The toys will be placed will be placed in drawers inside a cabinet. Inside the room, two brightly colored plastic Nerf dart guns and two handguns will be placed in separate drawers, as in previous research. The handguns will be modified so they cannot fire. Inside the magazine, the handguns contain no bullets. They do, however, contain a sensor that counts the number of times the trigger is depressed with sufficient force to discharge the weapon. This allows us to distinguish reliably the children who pull the trigger from those who only handle the gun. Parents will be asked to predict whether their child will handle the real gun and pull the trigger. The researcher and the parents will be able to watch the session via a monitor in a control room. A thorough debriefing will follow (see attachment). The investigators also have received letters of support from the Director of the School of Communication and from the Chief of Police (see attachments). The investigators predict the highest levels of playing with guns and firing them among participants who see a violent clip containing guns.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-12yrs, had not participated in study prior, was able to schedule participation with a known peer (8-12yo).

Exclusion Criteria:

* Younger than 8yo, older than 12yo, had participated in study prior, could not schedule participation with a known peer (8-12yo)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are considering making individual participant data available, but need to determine steps and appropriateness according to our institutional IRB board.

REFERENCES:
- [Derived] Chang JH, Bushman BJ. Effect of Exposure to Gun Violence in Video Games on Children's Dangerous Behavior With Real Guns: A Randomized Clinical Trial. JAMA Netw Open. 2019 May 3;2(5):e194319. doi: 10.1001/jamanetworkopen.2019.4319. PMID 31150072

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were both randomly assigned to condition (i.e. non-violent, sword, gun conditions) and to be either a player or watcher.
Groups:
- Experimental: Violence With Guns (Player): Participants in this condition will play a video game with violent content which includes guns.
  Video games and violence: Participants will be randomly assigned to play a video game which contains either (1) no violent content, (2) violent content with swords, or (3) violent content with guns. The game, rated E, is age appropriate and modded to include guns in the appropriate condition.
- Experimental: Violence With Guns (Watcher): Participants in this condition will watch a video game with violent content which includes guns.
  Video games and violence: Participants will be randomly assigned to play a video game which contains either (1) no violent content, (2) violent content with swords, or (3) violent content with guns. The game, rated E, is age appropriate and modded to include guns in the appropriate condition.
- Experimental: Violence Without Guns (Player): Participants in this condition will play a video game with violent content which does not include guns. Instead, the violence will include weapons such as swords.
  Video games and violence: Participants will be randomly assigned to play a video game which contains either (1) no violent content, (2) violent content with swords, or (3) violent content with guns. The game, rated E, is age appropriate and modded to include guns in the appropriate condition.
- Experimental: Violence Without Guns (Watcher); Control: No Violence (Watcher): Participants in this condition will watch a video game with violent content which does not include guns. Instead, the violence will include weapons such as swords.
  Video games and violence: Participants will be randomly assigned to play a video game which contains either (1) no violent content, (2) violent content with swords, or (3) violent content with guns. The game, rated E, is age appropriate and modded to include guns in the appropriate condition.
- Control: No Violence (Player): Participants in this condition will play a video game which contains no violent content or weapons.
  Video games and violence: Participants will be randomly assigned to play a video game which contains either (1) no violent content, (2) violent content with swords, or (3) violent content with guns. The game, rated E, is age appropriate and modded to include guns in the appropriate condition.
Period: Overall Study
Arm/Group | Experimental: Violence With Guns (Player) | Experimental: Violence With Guns (Watcher) | Experimental: Violence Without Guns (Player) | Experimental: Violence Without Guns (Watcher) | Control: No Violence (Player) | Control: No Violence (Watcher)
Started | 42 | 42 | 42 | 42 | 41 | 41
Eligible | 41 | 41 | 41 | 41 | 41 | 41
Outlier Elimination | 41 | 41 | 41 | 41 | 39 | 39
Found Handgun | 38 | 38 | 37 | 37 | 35 | 35
Completed | 38 | 38 | 37 | 37 | 35 | 35
Not Completed | 4 | 4 | 5 | 5 | 6 | 6

BASELINE CHARACTERISTICS:
Population: Children between the ages of 8 - 12, tested in pairs. Several children were excluded from the analysis, either for not meeting study criteria (n=4), for being identified as outliers (n=4), or for not finding the handguns (n=22). Figures here are after exclusions.
Groups:
- Control: No Violence (Watcher): Participants in this condition will watch a video game which contains no violent content or weapons.
  Video games and violence: Participants will be randomly assigned to play a video game which contains either (1) no violent content, (2) violent content with swords, or (3) violent content with guns. The game, rated E, is age appropriate and modded to include guns in the appropriate condition.
- Total: Total of all reporting groups
Arm/Group | Experimental: Violence With Guns (Player) | Experimental: Violence With Guns (Watcher) | Experimental: Violence Without Guns (Player) | Experimental: Violence Without Guns (Watcher) | Control: No Violence (Player) | Control: No Violence (Watcher) | Total
Number analyzed (Participants) | 38 | 38 | 37 | 37 | 35 | 35 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: NOTE: One parent or guardian did not provide this information on their child. This child was in the "No Violence (player)" condition. As such, measures for that condition were calculated with 34 instead of 35 participants.
  years
    number analyzed (Participants) | 38 | 38 | 37 | 37 | 34 | 35 | 219
    (all) | 9.66 (1.60) | 10.08 (1.50) | 9.97 (1.21) | 9.95 (1.41) | 9.88 (1.40) | 9.82 (1.36) | 9.94 (1.45)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This information was available for all 220 participants.
  Participants
    Female | 16 | 15 | 11 | 15 | 13 | 21 | 91
    Male | 22 | 23 | 26 | 22 | 22 | 14 | 129
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: NOTE: One parent or guardian did not provide this information on their child. This child was in the "No Violence (player)" condition. As such, measures for that condition were calculated with 34 instead of 35 participants.
  Participants
    White: number analyzed (Participants) | 38 | 38 | 37 | 37 | 34 | 35 | 219
    White | 28 | 28 | 28 | 26 | 26 | 27 | 163
    Black | 4 | 4 | 5 | 3 | 5 | 4 | 25
    Latino | 0 | 0 | 1 | 2 | 0 | 2 | 5
    Asian | 1 | 1 | 0 | 1 | 0 | 0 | 3
    Mixed race or other | 5 | 5 | 3 | 5 | 3 | 2 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 38 | 37 | 37 | 35 | 35 | 220

OUTCOME MEASURES:

1. Primary Outcome: Time Spent Holding Gun
Description: Time (in seconds) participant spent holding the real firearm during the play session
Time Frame: 20 minute play session
Population: NOTE: players and observers were collapsed into a single category for analysis
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Control: No Violence (Player) | Control: No Violence (Watcher) | Experimental: Violence Without Guns (Player) | Experimental: Violence Without Guns (Watcher) | Experimental: Violence With Guns (Player) | Experimental: Violence With Guns (Watcher)
Number analyzed (Participants) | 35 | 35 | 37 | 37 | 38 | 38
Seconds | 29.57 (15.28) | 21.14 (10.92) | 82.86 (25.79) | 48.62 (24.77) | 61.52 (17.77) | 68.40 (17.59)

2. Primary Outcome: Number of Trigger Pulls
Description: Number of times participant pulled trigger of real firearm during the play session
Time Frame: 20 minute play session
Population: NOTE: players and observers were collapsed into a single category for analysis
Measure: Mean (Standard Error); unit: Number of trigger pulls
Arm/Group | Control: No Violence (Player) | Control: No Violence (Watcher) | Experimental: Violence Without Guns (Player) | Experimental: Violence Without Guns (Watcher) | Experimental: Violence With Guns (Player) | Experimental: Violence With Guns (Watcher)
Number analyzed (Participants) | 35 | 35 | 37 | 37 | 38 | 38
Number of trigger pulls | 2.31 (1.60) | 1.97 (1.20) | 4.19 (1.74) | 2.22 (1.45) | 6.45 (2.60) | 8.79 (3.38)

3. Primary Outcome: Number of Trigger Pulls Aimed at Self or Other
Description: Trigger pulls while the firearm is aimed at the child holding the firearm or the other participant.
Time Frame: 20 minute play session
Population: NOTE: players and observers were collapsed into a single category for analysis
Measure: Mean (Standard Error); unit: Number of trigger pulls
Arm/Group | Control: No Violence | Control: No Violence (Watcher) | Experimental: Violence Without Guns | Experimental: Violence Without Guns (Watcher) | Experimental: Violence With Guns | Experimental: Violence With Guns (Watcher)
Number analyzed (Participants) | 35 | 35 | 37 | 37 | 38 | 38
Number of trigger pulls | 0.20 (0.20) | 0.09 (0.09) | 1.97 (1.22) | 0.84 (0.53) | 2.42 (1.17) | 3.68 (1.74)

ADVERSE EVENTS:
Time Frame: 1 week, as reported by parents in a follow-up email
Description: This study did not pose any serious risk to the participants.
Arm/Group | Experimental: Violence With Guns (Player) | Experimental: Violence With Guns (Watcher) | Experimental: Violence Without Guns (Player) | Experimental: Violence Without Guns (Watcher) | Control: No Violence (Player) | Control: No Violence (Watcher)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/37 | 0/37 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/37 | 0/37 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/37 | 0/37 | 0/35 | 0/35

LIMITATIONS AND CAVEATS:
Study setting was in a lab, i.e. not a natural setting, which may have caused subjects to be more likely to not think the guns are real. The game used was not very violent due to ethical reasons, so the effects may be larger with more violent games.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT03259139/Prot_SAP_000.pdf